CLINICAL TRIAL: NCT06784778
Title: A Prospective, Observational, Multicenter Clinical Performance Study to Evaluate IOpener®-Melanoma Test for Predicting Response to Combination or Mono Immunotherapy in Stage III or IV Cutaneous Melanoma Patients.
Brief Title: Observational Study of Patients With Advanced Melanoma (Skin Cancer) to Assess if IOpener®-Melanoma Test Can Predict Response to Immunotherapy.
Acronym: COMO
Status: Recruiting | Type: Observational
Sponsor: Pamgene International B.V. (Industry)
Collaborators: University Hospital Tuebingen (Other); lron Bridge GmbH (Unknown)
Responsible Party: Sponsor
Other Study IDs: IOpener®-melanoma COMO
Record Dates: First submitted 2025-01-06; First posted 2025-01-20 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-01

CONDITIONS: Melanoma Metastatic; Melanoma, Skin; Melanoma Stage III or IV; Melanoma Advanced
Keywords: melanoma; IOpener; immunotherapy; immune checkpoint inhibitor
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral Blood Mononuclear Cells (PBMCs) isolated from blood.
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (2):
- Standard of care anti-PD1 monotherapy: Patients receiving nivolumab or pembrolizumab.
  Interventions: Diagnostic Test: PBMC Kinase Activity Profile
- Standard of care combination therapy: Patients receiving ipilimumab plus nivolumab.
  Interventions: Diagnostic Test: PBMC Kinase Activity Profile

INTERVENTIONS:
Diagnostic Test: PBMC Kinase Activity Profile — Kinase activity profile will be correlated to the observed clinical outcome parameters (including survival and toxicity associated with the therapy) of standard of care treatments
  Other Names: IOpener-melanoma

SUMMARY:
The goal of this observational study is to assess whether the IOpener® melanoma test can assist treating physicians in deciding which therapy is most suitable for patients with skin cancer (advanced cutaneous melanoma). For this purpose it is evaluated how well the IOpener-melanoma test can predict the result of cancer treatment in the treatment groups (standard of care anti-PD1 mono-therapy and standard of care anti-PD1 + anti-CTLA-4 therapy).

Participants will be asked to provide blood sample for analysis using IOpener®-melanoma test. Patients will receive regular medical care, the test results will not be used to make any treatment decisions. The patients will visit the clinic for treatment administration and clinical evaluation as part of their regular medical care.

ELIGIBILITY:
Inclusion Criteria:

* First line treatment for unresectable stage III or IV cutaneous melanoma (according to AJCC version 8) with anti-PD1 monotherapy (nivolumab or pembrolizumab) or anti-PD1 + anti-CTL4A combination therapy (nivolumab and ipilimumab).
* Anticipated life expectancy exceeding 3 months.
* Aged 18 years or older and able to provide written informed consent.

Patients who have completed adjuvant treatment with anti-PD1 immunotherapy at least 6 months ago can be included.

Exclusion Criteria:

* Prior treatment for irresectable stage III or stage IV melanoma with BRAF/MEK inhibitors.
* Presence of progressive/symptomatic brain metastases at baseline.
* WHO performance score ≥ 2.
* Adjuvant treatment with anti-PD1 immunotherapy received within the last 6 months.
* Patients undergoing experimental treatments or therapies.
* Presence of any medical or other condition that in the opinion of the investigator(s) would preclude the participation in a clinical study.
* Unwillingness or inability to comply with study and follow-up procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced-stage melanoma who will receive standard-of-care treatment with immune checkpoint inhibitors (ICIs).
Sampling Method: Non-Probability Sample
Enrollment: 196 (Estimated)
Dates: Start 2024-07-12 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
12 months Progression Free Survival rate | From the enrollment to 12 months follow up.
  Predictive value of IOpener-melanoma for 1-year Progression Free Survival (PFS), i.e., proportion of patients without progressive disease (PD) ≥ 1 year, stratified according to treatment group and IOpener-melanoma test result.

SECONDARY OUTCOMES:
Disease Control Rate at 1 year | From enrollment to 12 months follow up.
  Disease Control Rate (DCR, "clinical benefit") at 1 year, based on Best Overall Response (BOR) according to RECIST 1.1.
Overall Response Rate (ORR) at 1 year | From enrollment to 12 months follow up.
  Overall Response Rate (ORR) at 1 year based on Best Overall Response (BOR) according to RECIST 1.1.
Progression Free Survival | From enrollment to month 24 follow up.
  Progression Free Survival
Overall Survival | From enrollment to month 24 follow up.
  Overall Survival

OTHER OUTCOMES:
Adverse events | From enrollment to month 24 follow up.
  Occurrence and type of adverse event or toxicity associated with standard of care.
Medical costs | From enrollment to month 24 follow up.
  Medical costs/medical care consumption associated with adverse events

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - Universitätsklinikum Tübingen, Tübingen, Baden-Wurttemberg
  - Heidelberg University Hospital, Heidelberg
  - LMU Klinikum, München